CLINICAL TRIAL: NCT03100786
Title: A Randomized Double Blind Placebo Controlled Non-inferiority Trial of Adjunctive Dexamethasone for the Treatment of HIV-uninfected Adults With Tuberculous Meningitis Stratified by Leukotriene A4 Hydrolase Genotype
Brief Title: Leukotriene A4 Hydrolase Stratified Trial of Adjunctive Corticosteroids for HIV-uninfected Adults With Tuberculous Meningitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam (Other); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27TB; 110179/Z/15/Z (Other Grant/Funding Number: The Wellcome Trust)
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis; Tuberculous Meningitis; Drug-Induced Liver Injury
Keywords: Tuberculosis; tuberculous meningitis; drug induced liver injury; dexamethasone; LTA4H; host genotype; personalized medicine
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Meningeal; Chemical and Drug Induced Liver Injury | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Active Comparator): standard anti-tuberculosis drugs plus dexamethasone for 6-8 weeks
  Interventions: Drug: Dexamethasone
- Identical placebo (Placebo Comparator): standard anti-tuberculosis drugs plus placebo for 6-8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Active treatment with dexamethasone from randomisation (IV followed by oral according to disease severity at the start of treatment): Dexamethasone for intravenous injection and dexamethasone for oral ingestion
  Arms: Dexamethasone
Other: Placebo — Treatment with matched placebo: Standard saline for intravenous injection and placebo oral tablets containing cellulose
  Arms: Identical placebo

SUMMARY:
The primary objective is to determine whether Leukotriene A4 hydrolase (LTA4H) genotype, defined at randomisation, determines dexamethasone's clinical effectiveness when added to the first 6-8 weeks of anti-tuberculosis treatment of TBM. The investigators will conduct a LTA4H genotype stratified, parallel group, randomised, double blind, placebo-controlled multi-centre Phase III non-inferiority trial evaluating dexamethasone versus placebo for 6-8 weeks in addition to standard anti-tuberculosis drugs.

The investigators will take a hybrid trial-design approach which assumes a modest harm of dexamethasone and aims to prove non-inferiority of placebo first but also allows claiming superiority of placebo in case dexamethasone causes substantial harm. Moreover, as it is possible that harm of dexamethasone only applies to the LTA4H CC genotype, the trial will allow dropping the CT group at an interim analysis but continue randomization of the CC group.

In making this assessment the investigators not only determine whether dexamethasone influences survival and the incidence of new neurological events (the primary endpoint), but also whether it influences disability assessed by the modified Rankin score 12 months after the start of treatment.

The secondary objective is to investigate alternative management strategies in a subset of patients who develop drug-induced liver injury that will enable the safe continuation of rifampicin and isoniazid therapy whenever possible.

DETAILED DESCRIPTION:
There is a longstanding hypothesis that death from TBM results from an excessive intracerebral inflammatory response. The corollary of this hypothesis has been that adjunctive anti-inflammatory treatment with corticosteroids (e.g. dexamethasone) improves survival, which has been demonstrated in predominantly HIV-uninfected individuals in a small number of trials. Yet how corticosteroids improve survival, and whether they do so in all patients, remain uncertain and is the focus of the LAST ACT trial.

Adjunctive dexamethasone might improve outcomes from TBM by controlling the early intracerebral inflammatory response, reducing cerebral oedema and intra-cranial pressure, and it may prevent the potentially life-threatening complications of hydrocephalus, infarction and tuberculoma formation. Despite the careful study of all participants enrolled into the last dexamethasone trial conducted in Vietnam, an anti-inflammatory effect linked to outcome was not found. An explanation for these puzzling findings was only forthcoming upon the subsequent discovery that a common functional promoter variant (C/T transition) in the gene encoding leukotriene A4 hydrolase (LTA4H), which determines the balance of pro- and anti-inflammatory eicosanoids, appeared to predict pre-treatment inflammatory phenotype and response to dexamethasone in HIV-uninfected participants.

In a retrospective study, analysing HIV-uninfected Vietnamese adults with TBM enrolled into the earlier randomized controlled trial of adjunctive dexamethasone, the investigators found that the survival benefit of dexamethasone was restricted to the hyper-inflammatory LTA4H TT-genotype patients, with possible harm suggested in the hypo-inflammatory CC-genotype patients. These preliminary findings suggested LTA4H genotype might be a critical determinant of inflammation and consequently of adjunctive anti-inflammatory treatment response.

Recently, the investigators have extended these original observations in a new cohort of 786 prospectively characterized Vietnamese adults with TBM, all of whom received corticosteroids. In this new cohort the investigators found that LTA4H genotype influences the survival of HIV-uninfected patients, but not those infected with HIV in patients receiving dexamethasone. TT-genotype patients were significantly more likely to survive than CC-genotype patients by both univariable and multivariable analysis, which confirms the previous findings.

The investigators now have two independent studies that suggest LTA4H influences pre-treatment inflammatory phenotype in HIV-uninfected Vietnamese adults and dexamethasone-induced survival. The investigators now want to conduct a practice-defining RCT that addresses the hypothesis that in HIV-uninfected adults with TBM, LTA4H genotype can be used to select those most likely to benefit from dexamethasone.

The data strongly suggest 'hyperinflammatory' LTA4H TT genotype patients with TBM benefit from dexamethasone. Therefore, these patients will be enrolled to the trial and followed-up for 12 months but will receive open label dexamethasone for the first 6-8 weeks of anti-tuberculosis treatment.

The data supports the hypothesis that adjunctive dexamethasone does not benefit, and may cause harm, when given to LTA4H CT or CC-genotype Vietnamese adults with TBM. Therefore, participants with these two genotypes will be randomised to receive 6-8 weeks of placebo or dexamethasone in addition to anti-tuberculosis drugs.

The primary objective is to determine whether LTA4H genotype, defined at randomisation, determines dexamethasone's clinical effectiveness when added to the first 6-8 weeks of anti-tuberculosis treatment of TBM. In making this assessment the investigators not only determine whether dexamethasone increases survival and reduces the incidence of new neurological events (the primary endpoint), but also whether it reduces disability assessed by the modified Rankin score 12 months after the start of treatment. The primary endpoint is death or new neurological event (defined as a fall in Glasgow coma score by ≥2 points for ≥2 days from the highest previously recorded Glasgow coma score (including baseline) or the onset of any of the following clinical adverse events: cerebellar symptoms, focal neurological signs, or new onset of seizures) during 12 months from randomisation.

The secondary objective is to investigate alternative management strategies in a subset of patients who develop drug-induced liver injury that will enable the safe continuation of rifampicin and isoniazid therapy whenever possible. The investigators will perform an open, randomised comparison of three management strategies with the aim of demonstrating which strategy results in the least interruption in R and H treatment. All patients enrolled in the trial will be eligible to take part in this study, with the exception of those known to have TBM caused by isoniazid resistant or MDR M. tuberculosis. Consent will be sought at enrolment, with an option given to patients to enrol in the main study, but not the 'drug-induced liver injury strategy study'.

Eligible patients will be randomised to one of three strategies:

1. Observe: measure transaminases, bilirubin, and INR every 3 days; do not change/stop anti-tuberculosis drugs unless transaminases rise to ≥10x normal, or total bilirubin rises >2.0mg/dl (>34 µmol/L), or INR >1.5 or symptoms of hepatitis worsen (nausea, vomiting, abdominal pain), in which case go to Strategy 3.
2. Stop Pyrazinamide (Z) alone. Observe, measuring transaminases, bilirubin, and INR every 3 days. If transaminases do not fall to < 5x ULN by day 5, or total bilirubin rises >2.0mg/dl (>34 µmol/L), or INR >1.5 or symptoms of hepatitis worsen at any time (nausea, vomiting, abdominal pain), go to Strategy 3.
3. Current standard of care (the current USA CDC guidelines): stop rifampicin (R), isoniazid (H) and Z immediately and add levofloxacin and an aminoglycoside to ethambutol. Restart R (at full dose) once transaminases are <2X ULN and no hepatitis symptoms. If no increase in transaminases after 7 days add isoniazid (at full dose) and stop levofloxacin and aminoglycoside. If transaminases remain normal on full dose R and H, Z was the likely cause and it should not be re-started and treatment duration should be extended to ≥12 months. If transaminases rise ≥ 5x ULN, or ≥3x ULN with symptoms, at any time after re-introduction of R and/or H the physician should stop R and/or H (depending on which was associated with the transaminase rise). If neither R or H can be used, treat with levofloxacin, an aminoglycoside and ethambutol. If R can be used, but not H, treat with R, levofloxacin and ethambutol. If H can be used, but not R, treat with H, levofloxacin and ethambutol.

The primary endpoint is the proportion of time in the 60 days following randomisation during which neither rifampicin nor isoniazid are given (or the subject is dead). For example, if RH is interrupted for 18 days and the participant dies 48 days after randomization, the endpoint will be 50% [(18+(60-48))/60]. Rifampicin and isoniazid are considered critical drugs in early TBM treatment; inability to use these agents (either through bacterial resistance or patient intolerance) is associated with poor outcome. The vast majority of interruptions are expected to be shorter than one month for strategy 3 (standard of care) but as management strategies 1 and 2 delay the time point of the interruption, a longer cut-off of 60 days was chosen.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* HIV-uninfected
* Clinical diagnosis of TBM (≥5 days of meningitis symptoms, and CSF abnormalities) and anti-tuberculosis chemotherapy either planned or started by the attending physician

Note: Published diagnostic criteria will be applied to all enrolled participants at the end of the study when all mycobacterial culture results are available. The criteria will sub-divide all cases into definite, probable and possible TBM, and those with an alternative diagnosis.

Exclusion Criteria:

* An additional brain infection (other than TBM) confirmed or suspected: positive CSF Gram or India Ink stain; positive blood or CSF Cryptococcal antigen test
* More than 6 consecutive days of two or more drugs active against M. tuberculosis immediately before screening
* More than 3 consecutive days of any type of orally or intravenously administered corticosteroid immediately before randomisation
* Dexamethasone considered mandatory for any reason by the attending physician
* Dexamethasone considered to be contraindicated for any reason by the attending physician
* Previously been randomised into the trial for a prior episode of TBM
* Lack of consent from the participant or family member (if the participant is incapacitated by the disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2024-03-09 (Actual)

PRIMARY OUTCOMES:
All-cause mortality or new neurological event | 12 months from randomisation
  The primary endpoint is all cause mortality or new neurological event (defined as a fall in Glasgow coma score by ≥2 points for ≥2 days from the highest previously recorded Glasgow coma score (including baseline) or the onset of any of the following clinical adverse events: cerebellar symptoms, focal neurological signs, or new onset of seizures) during 12 months from randomisation. Survivors without a new neurological event known to be alive at 12 months will be censored at that time-point and subjects who withdrew or were lost to follow-up before 12 months will be censored at the date they were last known to be alive.

SECONDARY OUTCOMES:
Overall survival until 12 months after randomization | 12 months after randomization
  Overall survival is defined as the time from randomization to death, during a follow-up period of 12 months. Survivors known to be alive at 12 months will be censored at that time-point and subjects who withdrew or were lost to follow-up before 12 months will be censored at the date they were last known to be alive.
Neurological disability at 12 months (modified Rankin score) | at 12 months
  Neurological disability will be assessed by the modified Rankin score on months 3, 6, 9, and 12 from randomisation. The main endpoint is the 12 month assessment and subjects who died before 12 months will be treated as having a score of 6 ('Dead')
Severe (grade 3 and 4) and serious adverse events by 12 months | by 12 months
  Comparison of the frequency of severe (grade 3&4) and serious adverse events, respectively, between treatment groups will form an important part of the study analysis.
Requirement for 'rescue' corticosteroids | during the 12 month follow-up
  Neurological complications occurring after the start of anti-tuberculosis chemotherapy for TBM are common. The cause varies, but includes hydrocephalus, infarcts, tuberculoma formation and hyponatraemia. If the symptoms are thought to be caused by tuberculomas, many doctors will re-start or increase the dose of corticosteroids. In this trial, any re-start or dose increase of corticosteroids during the 12 month follow-up will be defined as 'rescue' corticosteroids.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Thwaites, MD, Principal Investigator — University of Oxford, UK
Locations (3):
- Vietnam (3):
  - Hospital for Tropical Diseases, Ho Chi Minh City
  - Oxford University Clinical Research Unit, Ho Chi Minh City
  - Pham Ngoc Thach Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
The Oxford University Clinical Research Unit recognizes the ethical obligation to ensure that optimal use is made of the data and specimens that the investigators collect for the research and the value of sharing individual level data. The investigators aim to ensure that data generated from all the research are collected, curated, managed and shared in a way that maximizes their benefit. When sharing data the investigators have an obligation to ensure that the interests of research participants, researchers and other stakeholders are appropriately protected. The Oxford University Clinical Research Unit data sharing policy and the data request form outline the default procedures for data sharing.

REFERENCES:
- [Background] Thwaites GE, van Toorn R, Schoeman J. Tuberculous meningitis: more questions, still too few answers. Lancet Neurol. 2013 Oct;12(10):999-1010. doi: 10.1016/S1474-4422(13)70168-6. Epub 2013 Aug 23. PMID 23972913
- [Background] Kalita J, Misra UK. Outcome of tuberculous meningitis at 6 and 12 months: a multiple regression analysis. Int J Tuberc Lung Dis. 1999 Mar;3(3):261-5. PMID 10094329
- [Background] Thwaites GE, Duc Bang N, Huy Dung N, Thi Quy H, Thi Tuong Oanh D, Thi Cam Thoa N, Quang Hien N, Tri Thuc N, Ngoc Hai N, Thi Ngoc Lan N, Ngoc Lan N, Hong Duc N, Ngoc Tuan V, Huu Hiep C, Thi Hong Chau T, Phuong Mai P, Thi Dung N, Stepniewska K, Simmons CP, White NJ, Tinh Hien T, Farrar JJ. The influence of HIV infection on clinical presentation, response to treatment, and outcome in adults with Tuberculous meningitis. J Infect Dis. 2005 Dec 15;192(12):2134-41. doi: 10.1086/498220. Epub 2005 Nov 15. PMID 16288379
- [Background] STEWART SM. The bacteriological diagnosis of tuberculous meningitis. J Clin Pathol. 1953 Aug;6(3):241-2. doi: 10.1136/jcp.6.3.241. No abstract available. PMID 13084774
- [Background] Fallon RJ, Kennedy DH. Rapid diagnosis of tuberculous meningitis. J Infect. 1993 Mar;26(2):226. doi: 10.1016/0163-4453(93)93247-2. No abstract available. PMID 8473775
- [Background] Thwaites GE, Chau TT, Farrar JJ. Improving the bacteriological diagnosis of tuberculous meningitis. J Clin Microbiol. 2004 Jan;42(1):378-9. doi: 10.1128/JCM.42.1.378-379.2004. PMID 14715783
- [Background] Nhu NT, Heemskerk D, Thu do DA, Chau TT, Mai NT, Nghia HD, Loc PP, Ha DT, Merson L, Thinh TT, Day J, Chau Nv, Wolbers M, Farrar J, Caws M. Evaluation of GeneXpert MTB/RIF for diagnosis of tuberculous meningitis. J Clin Microbiol. 2014 Jan;52(1):226-33. doi: 10.1128/JCM.01834-13. Epub 2013 Nov 6. PMID 24197880
- [Background] Patel VB, Connolly C, Singh R, Lenders L, Matinyenya B, Theron G, Ndung'u T, Dheda K. Comparison of amplicor and GeneXpert MTB/RIF tests for diagnosis of tuberculous meningitis. J Clin Microbiol. 2014 Oct;52(10):3777-80. doi: 10.1128/JCM.01235-14. Epub 2014 Jul 23. PMID 25056328
- [Background] Thwaites G, Fisher M, Hemingway C, Scott G, Solomon T, Innes J; British Infection Society. British Infection Society guidelines for the diagnosis and treatment of tuberculosis of the central nervous system in adults and children. J Infect. 2009 Sep;59(3):167-87. doi: 10.1016/j.jinf.2009.06.011. Epub 2009 Jul 4. PMID 19643501
- [Background] Masur H, Brooks JT, Benson CA, Holmes KK, Pau AK, Kaplan JE; National Institutes of Health; Centers for Disease Control and Prevention; HIV Medicine Association of the Infectious Diseases Society of America. Prevention and treatment of opportunistic infections in HIV-infected adults and adolescents: Updated Guidelines from the Centers for Disease Control and Prevention, National Institutes of Health, and HIV Medicine Association of the Infectious Diseases Society of America. Clin Infect Dis. 2014 May;58(9):1308-11. doi: 10.1093/cid/ciu094. Epub 2014 Feb 27. PMID 24585567
- [Background] Thwaites GE. Advances in the diagnosis and treatment of tuberculous meningitis. Curr Opin Neurol. 2013 Jun;26(3):295-300. doi: 10.1097/WCO.0b013e3283602814. PMID 23493162
- [Background] Ellard GA, Humphries MJ, Allen BW. Cerebrospinal fluid drug concentrations and the treatment of tuberculous meningitis. Am Rev Respir Dis. 1993 Sep;148(3):650-5. doi: 10.1164/ajrccm/148.3.650. PMID 8368635
- [Background] Ruslami R, Ganiem AR, Dian S, Apriani L, Achmad TH, van der Ven AJ, Borm G, Aarnoutse RE, van Crevel R. Intensified regimen containing rifampicin and moxifloxacin for tuberculous meningitis: an open-label, randomised controlled phase 2 trial. Lancet Infect Dis. 2013 Jan;13(1):27-35. doi: 10.1016/S1473-3099(12)70264-5. Epub 2012 Oct 25. PMID 23103177
- [Background] Heemskerk AD, Bang ND, Mai NT, Chau TT, Phu NH, Loc PP, Chau NV, Hien TT, Dung NH, Lan NT, Lan NH, Lan NN, Phong le T, Vien NN, Hien NQ, Yen NT, Ha DT, Day JN, Caws M, Merson L, Thinh TT, Wolbers M, Thwaites GE, Farrar JJ. Intensified Antituberculosis Therapy in Adults with Tuberculous Meningitis. N Engl J Med. 2016 Jan 14;374(2):124-34. doi: 10.1056/NEJMoa1507062. PMID 26760084
- [Background] Tho DQ, Torok ME, Yen NT, Bang ND, Lan NT, Kiet VS, van Vinh Chau N, Dung NH, Day J, Farrar J, Wolbers M, Caws M. Influence of antituberculosis drug resistance and Mycobacterium tuberculosis lineage on outcome in HIV-associated tuberculous meningitis. Antimicrob Agents Chemother. 2012 Jun;56(6):3074-9. doi: 10.1128/AAC.00319-12. Epub 2012 Apr 2. PMID 22470117
- [Background] Thwaites GE, Lan NT, Dung NH, Quy HT, Oanh DT, Thoa NT, Hien NQ, Thuc NT, Hai NN, Bang ND, Lan NN, Duc NH, Tuan VN, Hiep CH, Chau TT, Mai PP, Dung NT, Stepniewska K, White NJ, Hien TT, Farrar JJ. Effect of antituberculosis drug resistance on response to treatment and outcome in adults with tuberculous meningitis. J Infect Dis. 2005 Jul 1;192(1):79-88. doi: 10.1086/430616. Epub 2005 May 20. PMID 15942897
- [Background] Seddon JA, Visser DH, Bartens M, Jordaan AM, Victor TC, van Furth AM, Schoeman JF, Schaaf HS. Impact of drug resistance on clinical outcome in children with tuberculous meningitis. Pediatr Infect Dis J. 2012 Jul;31(7):711-6. doi: 10.1097/INF.0b013e318253acf8. PMID 22411053
- [Background] Dass R, Nagaraj R, Murlidharan J, Singhi S. Hyponatraemia and hypovolemic shock with tuberculous meningitis. Indian J Pediatr. 2003 Dec;70(12):995-7. doi: 10.1007/BF02723828. PMID 14719791
- [Background] Figaji AA, Fieggen AG. The neurosurgical and acute care management of tuberculous meningitis: evidence and current practice. Tuberculosis (Edinb). 2010 Nov;90(6):393-400. doi: 10.1016/j.tube.2010.09.005. Epub 2010 Oct 20. PMID 20970381
- [Background] Celik U, Celik T, Tolunay O, Baspinar H, Komur M, Levent F. Cerebral salt wasting in tuberculous meningitis: Two cases and review of the literature. Case Report. Neuro Endocrinol Lett. 2015;36(4):306-10. PMID 26454484
- [Background] Schoeman J, Donald P, van Zyl L, Keet M, Wait J. Tuberculous hydrocephalus: comparison of different treatments with regard to ICP, ventricular size and clinical outcome. Dev Med Child Neurol. 1991 May;33(5):396-405. doi: 10.1111/j.1469-8749.1991.tb14899.x. PMID 2065826
- [Background] Chugh A, Husain M, Gupta RK, Ojha BK, Chandra A, Rastogi M. Surgical outcome of tuberculous meningitis hydrocephalus treated by endoscopic third ventriculostomy: prognostic factors and postoperative neuroimaging for functional assessment of ventriculostomy. J Neurosurg Pediatr. 2009 May;3(5):371-7. doi: 10.3171/2009.1.PEDS0947. PMID 19409015
- [Background] Thwaites GE, Macmullen-Price J, Tran TH, Pham PM, Nguyen TD, Simmons CP, White NJ, Tran TH, Summers D, Farrar JJ. Serial MRI to determine the effect of dexamethasone on the cerebral pathology of tuberculous meningitis: an observational study. Lancet Neurol. 2007 Mar;6(3):230-6. doi: 10.1016/S1474-4422(07)70034-0. PMID 17303529
- [Background] Sheu JJ, Hsu CY, Yuan RY, Yang CC. Clinical characteristics and treatment delay of cerebral infarction in tuberculous meningitis. Intern Med J. 2012 Mar;42(3):294-300. doi: 10.1111/j.1445-5994.2010.02256.x. Epub 2010 May 11. PMID 20492009
- [Background] Shukla R, Abbas A, Kumar P, Gupta RK, Jha S, Prasad KN. Evaluation of cerebral infarction in tuberculous meningitis by diffusion weighted imaging. J Infect. 2008 Oct;57(4):298-306. doi: 10.1016/j.jinf.2008.07.012. Epub 2008 Aug 28. PMID 18760486
- [Background] Springer P, Swanevelder S, van Toorn R, van Rensburg AJ, Schoeman J. Cerebral infarction and neurodevelopmental outcome in childhood tuberculous meningitis. Eur J Paediatr Neurol. 2009 Jul;13(4):343-9. doi: 10.1016/j.ejpn.2008.07.004. Epub 2008 Aug 30. PMID 18757219
- [Background] Koh SB, Kim BJ, Park MH, Yu SW, Park KW, Lee DH. Clinical and laboratory characteristics of cerebral infarction in tuberculous meningitis: a comparative study. J Clin Neurosci. 2007 Nov;14(11):1073-7. doi: 10.1016/j.jocn.2006.07.014. PMID 17954374
- [Background] Schoeman JF, Janse van Rensburg A, Laubscher JA, Springer P. The role of aspirin in childhood tuberculous meningitis. J Child Neurol. 2011 Aug;26(8):956-62. doi: 10.1177/0883073811398132. Epub 2011 May 31. PMID 21628697
- [Background] Misra UK, Kalita J, Nair PP. Role of aspirin in tuberculous meningitis: a randomized open label placebo controlled trial. J Neurol Sci. 2010 Jun 15;293(1-2):12-7. doi: 10.1016/j.jns.2010.03.025. Epub 2010 Apr 24. PMID 20421121
- [Background] Smith KU, Putz V. Feedback factors in steering and tracking behavior. J Appl Psychol. 1970 Apr;54(2):176-83. doi: 10.1037/h0028933. No abstract available. PMID 5496623
- [Background] Ramappa V, Aithal GP. Hepatotoxicity Related to Anti-tuberculosis Drugs: Mechanisms and Management. J Clin Exp Hepatol. 2013 Mar;3(1):37-49. doi: 10.1016/j.jceh.2012.12.001. Epub 2012 Dec 20. PMID 25755470
- [Background] Prasad K, Singh MB. Corticosteroids for managing tuberculous meningitis. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD002244. doi: 10.1002/14651858.CD002244.pub3. PMID 18254003
- [Background] Prasad K, Singh MB, Ryan H. Corticosteroids for managing tuberculous meningitis. Cochrane Database Syst Rev. 2016 Apr 28;4(4):CD002244. doi: 10.1002/14651858.CD002244.pub4. PMID 27121755
- [Background] Torok ME, Nguyen DB, Tran TH, Nguyen TB, Thwaites GE, Hoang TQ, Nguyen HD, Tran TH, Nguyen TC, Hoang HT, Wolbers M, Farrar JJ. Dexamethasone and long-term outcome of tuberculous meningitis in Vietnamese adults and adolescents. PLoS One. 2011;6(12):e27821. doi: 10.1371/journal.pone.0027821. Epub 2011 Dec 8. PMID 22174748
- [Background] Simmons CP, Thwaites GE, Quyen NT, Chau TT, Mai PP, Dung NT, Stepniewska K, White NJ, Hien TT, Farrar J. The clinical benefit of adjunctive dexamethasone in tuberculous meningitis is not associated with measurable attenuation of peripheral or local immune responses. J Immunol. 2005 Jul 1;175(1):579-90. doi: 10.4049/jimmunol.175.1.579. PMID 15972695
- [Background] Tobin DM, Roca FJ, Oh SF, McFarland R, Vickery TW, Ray JP, Ko DC, Zou Y, Bang ND, Chau TT, Vary JC, Hawn TR, Dunstan SJ, Farrar JJ, Thwaites GE, King MC, Serhan CN, Ramakrishnan L. Host genotype-specific therapies can optimize the inflammatory response to mycobacterial infections. Cell. 2012 Feb 3;148(3):434-46. doi: 10.1016/j.cell.2011.12.023. PMID 22304914
- [Background] Tobin DM, Vary JC Jr, Ray JP, Walsh GS, Dunstan SJ, Bang ND, Hagge DA, Khadge S, King MC, Hawn TR, Moens CB, Ramakrishnan L. The lta4h locus modulates susceptibility to mycobacterial infection in zebrafish and humans. Cell. 2010 Mar 5;140(5):717-30. doi: 10.1016/j.cell.2010.02.013. PMID 20211140
- [Background] Torok ME, Yen NT, Chau TT, Mai NT, Phu NH, Mai PP, Dung NT, Chau NV, Bang ND, Tien NA, Minh NH, Hien NQ, Thai PV, Dong DT, Anh DT, Thoa NT, Hai NN, Lan NN, Lan NT, Quy HT, Dung NH, Hien TT, Chinh NT, Simmons CP, de Jong M, Wolbers M, Farrar JJ. Timing of initiation of antiretroviral therapy in human immunodeficiency virus (HIV)--associated tuberculous meningitis. Clin Infect Dis. 2011 Jun;52(11):1374-83. doi: 10.1093/cid/cir230. PMID 21596680
- [Background] Thwaites GE, Bhavnani SM, Chau TT, Hammel JP, Torok ME, Van Wart SA, Mai PP, Reynolds DK, Caws M, Dung NT, Hien TT, Kulawy R, Farrar J, Ambrose PG. Randomized pharmacokinetic and pharmacodynamic comparison of fluoroquinolones for tuberculous meningitis. Antimicrob Agents Chemother. 2011 Jul;55(7):3244-53. doi: 10.1128/AAC.00064-11. Epub 2011 Apr 18. PMID 21502621
- [Background] Freidlin B, Korn EL, George SL, Gray R. Randomized clinical trial design for assessing noninferiority when superiority is expected. J Clin Oncol. 2007 Nov 1;25(31):5019-23. doi: 10.1200/JCO.2007.11.8711. PMID 17971602
- [Background] Spiessens B, Debois M. Adjusted significance levels for subgroup analyses in clinical trials. Contemp Clin Trials. 2010 Nov;31(6):647-56. doi: 10.1016/j.cct.2010.08.011. Epub 2010 Sep 9. PMID 20832503
- [Background] Lokhnygina Y, Helterbrand JD. Cox regression methods for two-stage randomization designs. Biometrics. 2007 Jun;63(2):422-8. doi: 10.1111/j.1541-0420.2007.00707.x. Epub 2007 Apr 9. PMID 17425633
- [Background] Saukkonen JJ, Cohn DL, Jasmer RM, Schenker S, Jereb JA, Nolan CM, Peloquin CA, Gordin FM, Nunes D, Strader DB, Bernardo J, Venkataramanan R, Sterling TR; ATS (American Thoracic Society) Hepatotoxicity of Antituberculosis Therapy Subcommittee. An official ATS statement: hepatotoxicity of antituberculosis therapy. Am J Respir Crit Care Med. 2006 Oct 15;174(8):935-52. doi: 10.1164/rccm.200510-1666ST. PMID 17021358
- [Background] Devarbhavi H, Singh R, Patil M, Sheth K, Adarsh CK, Balaraju G. Outcome and determinants of mortality in 269 patients with combination anti-tuberculosis drug-induced liver injury. J Gastroenterol Hepatol. 2013 Jan;28(1):161-7. doi: 10.1111/j.1440-1746.2012.07279.x. PMID 23020522
- [Background] Pukenyte E, Lescure FX, Rey D, Rabaud C, Hoen B, Chavanet P, Laiskonis AP, Schmit JL, May T, Mouton Y, Yazdanpanah Y. Incidence of and risk factors for severe liver toxicity in HIV-infected patients on anti-tuberculosis treatment. Int J Tuberc Lung Dis. 2007 Jan;11(1):78-84. PMID 17217134
- [Background] Sharma SK, Singla R, Sarda P, Mohan A, Makharia G, Jayaswal A, Sreenivas V, Singh S. Safety of 3 different reintroduction regimens of antituberculosis drugs after development of antituberculosis treatment-induced hepatotoxicity. Clin Infect Dis. 2010 Mar 15;50(6):833-9. doi: 10.1086/650576. PMID 20156055
- [Background] Tahaoglu K, Atac G, Sevim T, Tarun T, Yazicioglu O, Horzum G, Gemci I, Ongel A, Kapakli N, Aksoy E. The management of anti-tuberculosis drug-induced hepatotoxicity. Int J Tuberc Lung Dis. 2001 Jan;5(1):65-9. PMID 11263519
- [Background] Lenaerts A, Barry CE 3rd, Dartois V. Heterogeneity in tuberculosis pathology, microenvironments and therapeutic responses. Immunol Rev. 2015 Mar;264(1):288-307. doi: 10.1111/imr.12252. PMID 25703567
- [Background] Roca FJ, Ramakrishnan L. TNF dually mediates resistance and susceptibility to mycobacteria via mitochondrial reactive oxygen species. Cell. 2013 Apr 25;153(3):521-34. doi: 10.1016/j.cell.2013.03.022. Epub 2013 Apr 11. PMID 23582643
- [Background] Naranbhai V, Moodley D, Chipato T, Stranix-Chibanda L, Nakabaiito C, Kamateeka M, Musoke P, Manji K, George K, Emel LM, Richardson P, Andrew P, Fowler M, Fletcher H, McShane H, Coovadia HM, Hill AV; HPTN 046 Protocol Team. The association between the ratio of monocytes: lymphocytes and risk of tuberculosis among HIV-infected postpartum women. J Acquir Immune Defic Syndr. 2014 Dec 15;67(5):573-5. doi: 10.1097/QAI.0000000000000353. PMID 25247435
- [Background] Naranbhai V, Kim S, Fletcher H, Cotton MF, Violari A, Mitchell C, Nachman S, McSherry G, McShane H, Hill AV, Madhi SA. The association between the ratio of monocytes:lymphocytes at age 3 months and risk of tuberculosis (TB) in the first two years of life. BMC Med. 2014 Jul 17;12:120. doi: 10.1186/s12916-014-0120-7. PMID 25034889
- [Background] Naranbhai V, Hill AV, Abdool Karim SS, Naidoo K, Abdool Karim Q, Warimwe GM, McShane H, Fletcher H. Ratio of monocytes to lymphocytes in peripheral blood identifies adults at risk of incident tuberculosis among HIV-infected adults initiating antiretroviral therapy. J Infect Dis. 2014 Feb 15;209(4):500-9. doi: 10.1093/infdis/jit494. Epub 2013 Sep 16. PMID 24041796
- [Background] Sharma SK, Balamurugan A, Saha PK, Pandey RM, Mehra NK. Evaluation of clinical and immunogenetic risk factors for the development of hepatotoxicity during antituberculosis treatment. Am J Respir Crit Care Med. 2002 Oct 1;166(7):916-9. doi: 10.1164/rccm.2108091. PMID 12359646
- [Background] Dooley KE, Chaisson RE. Tuberculosis and diabetes mellitus: convergence of two epidemics. Lancet Infect Dis. 2009 Dec;9(12):737-46. doi: 10.1016/S1473-3099(09)70282-8. PMID 19926034
- [Background] Pizzol D, Di Gennaro F, Chhaganlal KD, Fabrizio C, Monno L, Putoto G, Saracino A. Tuberculosis and diabetes: current state and future perspectives. Trop Med Int Health. 2016 Jun;21(6):694-702. doi: 10.1111/tmi.12704. Epub 2016 May 18. PMID 27102229
- [Background] Salgame P, Yap GS, Gause WC. Effect of helminth-induced immunity on infections with microbial pathogens. Nat Immunol. 2013 Nov;14(11):1118-1126. doi: 10.1038/ni.2736. PMID 24145791
- [Background] George PJ, Pavan Kumar N, Jaganathan J, Dolla C, Kumaran P, Nair D, Banurekha VV, Shen K, Nutman TB, Babu S. Modulation of pro- and anti-inflammatory cytokines in active and latent tuberculosis by coexistent Strongyloides stercoralis infection. Tuberculosis (Edinb). 2015 Dec;95(6):822-828. doi: 10.1016/j.tube.2015.09.009. Epub 2015 Oct 8. PMID 26542223
- [Background] Hutchings S, Bisset L, Cantillon L, Keating-Brown P, Jeffreys S, Muzvidziwa C, Richmond E, Rees P. Nurse-delivered focused echocardiography to determine intravascular volume status in a deployed maritime critical care unit. J R Nav Med Serv. 2015;101(2):124-8. PMID 26867411
- [Background] Marik PE. Techniques for assessment of intravascular volume in critically ill patients. J Intensive Care Med. 2009 Sep-Oct;24(5):329-37. doi: 10.1177/0885066609340640. PMID 19648183
- [Background] Komut E, Kozaci N, Sonmez BM, Yilmaz F, Komut S, Yildirim ZN, Beydilli I, Yel C. Bedside sonographic measurement of optic nerve sheath diameter as a predictor of intracranial pressure in ED. Am J Emerg Med. 2016 Jun;34(6):963-7. doi: 10.1016/j.ajem.2016.02.012. Epub 2016 Feb 12. PMID 26944107
- [Background] Aduayi OS, Asaleye CM, Adetiloye VA, Komolafe EO, Aduayi VA. Optic nerve sonography: A noninvasive means of detecting raised intracranial pressure in a resource-limited setting. J Neurosci Rural Pract. 2015 Oct-Dec;6(4):563-7. doi: 10.4103/0976-3147.165347. PMID 26752428
- [Background] Magnusson BP, Turnbull BW. Group sequential enrichment design incorporating subgroup selection. Stat Med. 2013 Jul 20;32(16):2695-714. doi: 10.1002/sim.5738. Epub 2013 Jan 13. PMID 23315698
- [Derived] Donovan J, Duc Bang N, Dong HKT, Ho DTN, Nguyen TAT, Nguyen TTH, Lam HBN, Phung VKN, Nguyen TT, Nguyen HHH, Pham KNO, Do DAT, Nguyen TMT, Dang TMH, Nguyen HL, Nguyen VVC, Hoang TH, Tran DD, Phung KL, Ramakrishnan L, Le THN, Nguyen TTT, Wolbers M, Kestelyn E, Geskus RB, Nguyen HP, Thwaites GE. Genotype-stratified adjunctive dexamethasone for tuberculous meningitis in HIV-negative adults: a randomized controlled phase 3 trial. Nat Med. 2026 Jan 15. doi: 10.1038/s41591-025-04138-z. Online ahead of print. PMID 41540106
- [Derived] Donovan J, Oanh PKN, Dobbs N, Phu NH, Nghia HDT, Summers D, Thuong NTT, Thwaites GE; Vietnam ICU Translational Applications Laboratory (VITAL) Investigators. Optic Nerve Sheath Ultrasound for the Detection and Monitoring of Raised Intracranial Pressure in Tuberculous Meningitis. Clin Infect Dis. 2021 Nov 2;73(9):e3536-e3544. doi: 10.1093/cid/ciaa1823. PMID 33283229